CLINICAL TRIAL: NCT07096492
Title: Comparison of the Effects of Strength and Plyometric Training in 50-Meter Swimming
Brief Title: Strength and Plyometric Training in Swimming
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Çiçek Günday, Asst. Prof., Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07032025
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Sport Performance; Biomechanics; Plyometric Exercises; Strength Training Effects; Swimming
Keywords: Performance; Speed; Power; Biomechanics; Youth Swimmers
MeSH Terms: interventions — Plyometric Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric Group (Experimental)
  Interventions: Other: Standard Swimming Training; Other: Plyometric Training
- Strength Group (Experimental)
  Interventions: Other: Standard Swimming Training; Other: Strength Training

INTERVENTIONS:
Other: Standard Swimming Training — Warm-Up: 1500 meters. Main set: 2000-3000 meters. Post-set: 1000 meters. Cool-Down: 200-400 meters.
Other: Plyometric Training — The plyometric training intervention will focus on developing explosive power and reaction speed through various jumping and landing exercises. Progressive overload principles will be applied, with progression achieved through increasing sets and intensity. Plyometric exercises will be performed twice a week, similar to the strength group, and will begin with 3 sets of 3 repetitions in the first week. As the body adapts to the exercises, one additional set will be added each week until the third week, which will conclude with 5 sets. In the fourth week, a deload will be incorporated with 2 sets to allow for recovery. After the deload week, intensity will increase, either by performing exercises faster or exerting maximum effort during each repetition. Upper-body exercises will include the medicine ball slam, sitting medicine ball side passes, and medicine ball chest passes, focusing on explosive upper body movements. Lower-body exercises will consist of standing long jumps, partner med
  Arms: Plyometric Group
Other: Strength Training — The strength training intervention was designed to supplement standard swim training with a structured, full-body resistance program aimed at enhancing muscular strength and swimming biomechanics through progressive overload. Participants in the strength group engaged in two sessions per week for each major muscle group. Training commenced with 3 sets of 8 repetitions per exercise during the first week, with weekly increases in training volume until the third week (5 sets), followed by a deload week (3 sets) to promote recovery. The subsequent four weeks maintained a consistent 5-set structure, with progression achieved through incremental increases in load. Each session began with lower-body exercises to prioritize large muscle group activation and maximize session efficiency. Lower-body exercises included dumbbell goblet squats, step-ups, Romanian deadlifts, TRX hamstring curls, and calf raises, while upper-body work featured push-ups, TRX rows, dumbbell rows, and dumbbell shoulder p
  Arms: Strength Group

SUMMARY:
A total of 18 participants are planned to be included in the study. Participants will be randomly assigned into two groups in the order of their arrival. One group will perform strength exercises in addition to standard swim training (strength group), while the other group will perform plyometric exercises in addition to standard swim training (plyometric group). Both groups will participate in two training sessions per week for a duration of 8 weeks. The 50m sprint biomechanics, stroke frequency, or overall performance will be evaluated before and after the intervention.

DETAILED DESCRIPTION:
In sprint swimming events such as the 50-meter race, the ability to generate explosive power and maintain efficient biomechanics is critical for achieving peak performance. Plyometric training, particularly progressive bounding and long jump exercises, has been shown to effectively enhance the kinetic and kinematic parameters essential for swimming starts. This form of training plays a key role in sprint events that demand rapid propulsion, as it conditions the neuromuscular system to produce power quickly. As such, plyometric exercises directly contribute to improved initial push-off phases and overall sprint performance in short-distance swimming.

Similarly, strength training has a significant role in improving stroke length and stroke frequency. Low-volume, high-speed, and high-force strength training programs are particularly effective in transferring gains to swimming-specific mechanics. These improvements enhance stroke efficiency and power output, resulting in improved performance outcomes. In young swimmers, land-based strength and conditioning programs have demonstrated improvements in biomechanics, enabling swimmers to maintain higher speeds over 50 meters with minimal energy loss and more powerful strokes.

Collectively, these findings suggest that integrating plyometric and strength training into the training programs of young swimmers may yield beneficial effects on sprint biomechanics and overall performance. The current study aims to investigate the comparative effects of these two training modalities-plyometric and strength training-on 50-meter sprint performance and biomechanics in young swimmers. The results are expected to offer valuable insights into optimal conditioning strategies that support athletic development in competitive swimming.

Hypotheses:

Null Hypothesis (H₀): There is no significant difference in 50-meter sprint biomechanics, stroke frequency, or overall performance between young swimmers who undergo plyometric training in addition to swim training and those who undergo strength training in addition to swim training.

Alternative Hypothesis (H₁): There is a significant difference in 50-meter sprint biomechanics, stroke frequency, or overall performance between young swimmers who undergo plyometric training in addition to swim training and those who undergo strength training in addition to swim training.

Objectives:

To determine the chronic effects of plyometric training, in addition to regular swim training, on sprint biomechanics in young swimmers.

To evaluate the effects of strength training, in addition to regular swim training, on sprint biomechanics in young swimmers.

To compare developments in stroke frequency between the plyometric and strength training groups.

To examine the overall changes in 50-meter sprint performance in both training groups over the eight-week training period.

ELIGIBILITY:
Inclusion Criteria Being between 10 and 17 years old, Having at least 3 years of competitive experience, Having participated in at least one Qualifying Standards competition before, Being willing to participate in the study, Obtained parental consent.

Exclusion Criteria:

Presence of a health condition requiring regular medical check-ups (e.g., cardiovascular, respiratory, or musculoskeletal disorders).

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
50m Sprint Time (Overall Performance) | Through study completion, an average of 12 months
  The 50m sprint time is used as a direct measure of swimming performance and is evaluated both in freestyle and in the swimmer's primary stroke. This test is conducted before and after the 8-week training intervention using a stopwatch and high-resolution video equipment. Time splits are also recorded for the 15m and 25m marks to assess acceleration and speed maintenance phases. This measure provides a clear indication of whether the intervention (strength or plyometric training) leads to improved sprint capacity in competitive youth swimmers.
Sprint biomechanics and stroke frequency | Through study completion, an average of 12 months
  Biomechanics are assessed through underwater and above-water video analysis to evaluate body alignment, stroke path, and coordination. Stroke frequency, calculated from the same footage by timing three full stroke cycles, reflects how quickly a swimmer completes strokes. Together, these measures reveal whether performance gains stem from technical improvements, faster turnover, or more effective propulsion.

SECONDARY OUTCOMES:
Upper and Lower Body Muscle Strength | Through study completion, an average of 12 months
  Muscle strength is assessed using a Lafayette Hand-Held Dynamometer, which measures isometric force output in key joints (e.g., shoulder, hip, knee) for both upper and lower limbs. Each movement is tested in a standardized position, with three trials averaged per joint action. This outcome helps determine how much the dryland training programs contribute to the development of raw muscular strength, which is a foundational quality for explosive swimming movements.
Lower Body Explosive Power (Standing Long Jump Test) | Through study completion, an average of 12 months
  This test evaluates leg power through horizontal jump distance. Participants perform the test by bending their knees and using their arms to generate maximum forward momentum. The longest of several attempts is recorded as the final result. This test is especially relevant for assessing the effectiveness of the plyometric training group, as it reflects improvements in explosive leg power, which is critical for starts and turns in sprint swimming.

CONTACTS AND LOCATIONS:
Locations (1):
- Beylikdüzü Yüzme Kulübü, Istanbul, Beylikdüzü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes